CLINICAL TRIAL: NCT02854774
Title: Neural Mechanisms of Muscle Control in Individuals With Knee Pain
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No additional funding is available to continue this pilot study at this time.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jason Kutch, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-16-00038
Record Dates: First submitted 2016-06-07; First posted 2016-08-03 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee muscle activation/strengthening (Active Comparator): 4 weeks of exercises focused on activation and strengthening of knee extensor muscles.
  Interventions: Behavioral: Muscle activation exercises
- Hip muscle activation/strengthening (Active Comparator): 4 weeks of exercises focused on activation and strengthening of hip extensor muscles.
  Interventions: Behavioral: Muscle activation exercises

INTERVENTIONS:
Behavioral: Muscle activation exercises — Activation of either muscles activating the knee or hip.

SUMMARY:
This is a randomized controlled trial of knee muscle versus hip muscle strengthening for Patellofemoral Pain Syndrome.

DETAILED DESCRIPTION:
Rationale: Two prior randomized controlled trials (RCT) have highlighted the importance of hip muscle activation and strengthening as a treatment strategy for patellofemoral pain (Khayambashi, 2014; Khayambashi, 2012). Here, we propose a pilot study to acquire preliminary data to power a larger study to reveal the neural mechanism underlying the effectiveness of this intervention to promote its evidence-based incorporation into clinical practice.

Intervention: 4 weeks of quadriceps muscle versus 4 weeks of hip strengthening exercises.

Purpose: To determine changes in brain functional connectivity related to pain reduction induced by the strengthening exercises.

Study population: Males and females with a history of unilateral knee pain.

Methodology: Functional magnetic resonance imaging (fMRI) will be used to quantify functional connectivity of brain regions related to hip muscle activation. Functional connectivity will be quantified before (pre) and after (post) 4 weeks of quadricep or hip muscle strengthening exercises.

Arms: As above, there are 2 arms. 4 weeks of quadriceps strengthening exercises (Arm 1) versus 4 weeks of hip strengthening exercises (Arm 2).

Outcomes: At the pre and post-intervention sessions in each participant, we will quantify the brain functional connectivity between hip muscle motor cortex and the 1) thalamus, 2) basal ganglia, and 3) insula, and 4) the periaqueductal gray. We will also quantify self-report of pain and biomechanical function of the knee and hip.

Follow-up: A six month follow-up is planned for this pilot study.

Analysis Plan and Statistics: Functional connectivity of hip muscle motor cortex will be extracted using standard statistical software for brain mapping. A repeated measures ANOVA will be used to assess change in functional connectivity in the hip and knee group. Pain decreases in the both groups will be quantified and reported.

ELIGIBILITY:
Inclusion Criteria:

1. Pain located specifically around the patellofemoral articulation (vague or localized).
2. Readily reproducible pain (3 out of 10 on a visual analog scale) with at least 2 of the following functional activities commonly associated with PFP: stair ascent or descent, squatting, kneeling, prolonged sitting, or isometric quadriceps contraction.
3. Reports of pain greater than 3 months duration.

Exclusion Criteria:

1. Previous history of knee surgery.
2. History of traumatic patellar dislocation.
3. Neurological involvement that would influence gait.
4. Contraindications to MR imaging: implanted electronic devices (i.e. pacemaker), or metallic implants (i.e. aneurysm clips, fixation screws).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
Pain reduction measured using a visual analog scale (VAS) for knee pain | 4 weeks and 6 months
  Compared to baseline

SECONDARY OUTCOMES:
Brain function measured using fMRI | 4 weeks
  Compared to baseline
Muscle activation assessed with electromyographic (EMG) recordings | 4 weeks
  Activation of knee and hip muscles
Knee kinematics assessed with 3-dimensional motion capture | 4 weeks
  Body movement during a jumping task

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khayambashi K, Mohammadkhani Z, Ghaznavi K, Lyle MA, Powers CM. The effects of isolated hip abductor and external rotator muscle strengthening on pain, health status, and hip strength in females with patellofemoral pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):22-9. doi: 10.2519/jospt.2012.3704. Epub 2011 Oct 25. PMID 22027216
- [Result] Khayambashi K, Fallah A, Movahedi A, Bagwell J, Powers C. Posterolateral hip muscle strengthening versus quadriceps strengthening for patellofemoral pain: a comparative control trial. Arch Phys Med Rehabil. 2014 May;95(5):900-7. doi: 10.1016/j.apmr.2013.12.022. Epub 2014 Jan 16. PMID 24440362